CLINICAL TRIAL: NCT00983021
Title: A Trial to Test for Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NN9068 and Compared With NN1250 and NN2211 in Healthy Subjects
Brief Title: Safety and Tolerability of NN9068 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9068-3632; 2009-011269-95 (EudraCT Number); U1111-1111-8859 (Other: WHO)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — IDegLira; insulin degludec; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental)
  Interventions: Drug: insulin degludec/liraglutide; Drug: placebo
- B (Experimental)
  Interventions: Drug: insulin degludec; Drug: placebo
- C (Active Comparator)
  Interventions: Drug: liraglutide; Drug: placebo
- D (Experimental)
  Interventions: Drug: insulin degludec; Drug: liraglutide

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Single, simultaneous dose of NN9068, injected s.c. (under the skin)
  Other Names: NN9068
  Arms: A
Drug: insulin degludec — Single, simultaneous dose of NN1250, injected s.c. (under the skin)
  Other Names: NN1250
  Arms: B; D
Drug: liraglutide — Single, simultaneous dose of NN2211, injected s.c. (under the skin)
  Other Names: NN2211
  Arms: C; D
Drug: placebo — Single, simultaneous dose of placebo, injected s.c. (under the skin)
  Arms: A; B; C

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the safety, tolerability, level of drug exposure and effect of NN9068.

The trial participants will be randomised to 4 different treatments in trial, receiving trial products in a pre-defined order.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, who are considered to be generally healthy, based on an assessment of medical history, physical examination, and clinical laboratory data, as judged by the Investigator.
* Body mass index (BMI) between 18.0 and 27.0 kg/m2 (both inclusive)
* Body weight between 60 kg and 90 kg (both inclusive)

Exclusion Criteria:

* Subjects with a history of or presence of cancer, diabetes, or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders that might have impact on the current trial, as judged by the Investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events, number and severity of local tolerability issues at the injection site, number and severity of hypoglycaemic episodes | assessed 0-96 hours after trial product administration

SECONDARY OUTCOMES:
The area under the NN2211 concentration-time curve after single-dose | assessed 0-72 hours after trial product administration
The area under the NN1250 concentration-time curve after single-dose | assessed 0-96 hours after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Kapitza C, Bode B, Ingwersen SH, Jacobsen LV, Poulsen P. Preserved pharmacokinetic exposure and distinct glycemic effects of insulin degludec and liraglutide in IDegLira, a fixed-ratio combination therapy. J Clin Pharmacol. 2015 Dec;55(12):1369-77. doi: 10.1002/jcph.549. Epub 2015 Jul 14. PMID 25998481
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com